CLINICAL TRIAL: NCT03736863
Title: A Phase II Exploratory Clinical Trial of Multiple Drug Combinations in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FQX-001/MA-EC-II-002/CAP 02
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CohortA：Apatinib+SHR-1210（Camrelizumab） (Experimental): Apatinib+SHR-1210（Camrelizumab）for ESCC who progressed or were intolerant to first-line systemic chemotherapy
  Interventions: Drug: Apatinib+ SHR-1210（Camrelizumab）
- CohortB：Apatinib+SHR-1210（Camrelizumab） (Experimental): Apatinib+SHR-1210（Camrelizumab）for ESCC who have failed prior immune checkpoint inhibitor therapies
  Interventions: Drug: Apatinib+ SHR-1210（Camrelizumab）
- CohortC：Apatinib+SHR-1316（Adebrelimab） (Experimental): Apatinib+SHR-1316（Adebrelimab）for ESCC who have failed prior immune checkpoint inhibitor therapies
  Interventions: Drug: Apatinib+ SHR-1316（Adebrelimab）
- CohortD：SHR-1316（Adebrelimab）+SHR-A2009 (Experimental): SHR-1316 was administered intravenously, 1200mg, Q3W; SHR-A2009 8mg/kg, iv, Q3W, for ESCC who have failed prior immune checkpoint inhibitor therapies.
  Interventions: Drug: SHR-1316（Adebrelimab）+SHR-A2009

INTERVENTIONS:
Drug: Apatinib+ SHR-1210（Camrelizumab） — Apatinib 250mg, q.d.po+SHR-1210（Camrelizumab）200 mg，Intravenous injection，q2W
  Arms: CohortA：Apatinib+SHR-1210（Camrelizumab）; CohortB：Apatinib+SHR-1210（Camrelizumab）
Drug: Apatinib+ SHR-1316（Adebrelimab） — Apatinib 250mg, q.d.po+SHR-1316（Adebrelimab） 1200 mg，Intravenous injection，q2W
  Arms: CohortC：Apatinib+SHR-1316（Adebrelimab）
Drug: SHR-1316（Adebrelimab）+SHR-A2009 — SHR-1316 was administered intravenously, 1200mg, Q3W; SHR-A2009 8mg/kg, iv, Q3W,
  Arms: CohortD：SHR-1316（Adebrelimab）+SHR-A2009

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of multiple drug combinations in the treatment of advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Immunotherapy has been widely used in patients with advanced esophageal cancer. Immunochemotherapy has become the standard treatment for advanced esophageal squamous cell carcinoma. The common second-line standard treatment is immunotherapy or chemotherapy, but that are established according to the medical evidence after the progression of chemotherapy, the preferred treatment plan after immuno-resistance needs to be explored. The purpose of this study was to explore the efficacy and safety of different drug combinations in patients with advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, males or females;
2. Histologically or cytologically confirmed as ESCC, locally advanced and unresectable, with local recurrence (local lymph node metastases) or distant metastases;
3. First-line patients who progressed or were intolerant after chemotherapy (cohort A) or immumotherapy (other cohorts). Concurrent chemoradiotherapy with postoperative recurrence or metastasis is considered as first-line treatment. For radical concurrent chemoradiotherapy, neoadjuvant/adjuvant therapy (chemotherapy or chemoradiotherapy), if disease progression occurs during treatment or within 6 months after stopping treatment, it should be counted as first-line treatment failure;
4. The best overall response of first-line immunotherapy is CR, PR or SD, and PFS ≥ 3 months;
5. According to the Response Evaluation Criteria In Solid Tumour (RECIST 1.1), there is at least one measurable lesion, which has not received any local treatment, such as radiotherapy (if the lesion within the region of the previous radiotherapy is confirmed to progress and satisfies RECIST1.1, it can be also selected as the target lesion) ;
6. Tissue samples should be provided for biomarker analysis. The newly harvested tissues are preferred. If the newly harvested tissues are not available, 5-8 archival paraffin sections (5 um thick) can be provided;
7. ECOG: 0~1;
8. Expected survival time ≥ 12 weeks;
9. Adequate function of major organs defined as:(1) Routine blood test: a. HB ≥ 90 g/L; b. ANC ≥ 1.5 × 109/L; c. PLT ≥ 80 × 109/L;(2) Biochemical test: a. ALB ≥ 30 g/L; b. ALT and AST ≤ 2.5 ULN; if there is no liver metastasis, ALT and AST ≤ 5 ULN; c. TBIL ≤ 1.5ULN; d. Plasma Cr ≤ 1.5 ULN or creatinine clearance rate (CCr) ≥ 60 mL/min;
10. Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).
11. Women of childbearing age should consent to take contraception measures during the study period and within 6 months after the end of the study (eg., intrauterine device, oral contraceptive pills or condoms). The subjects must be negative for the serum or urine pregnancy test within 7 days before the recruitment. The female subjects must be non-lactating women. Males should consent to take contraception measures during the study period and within 6 months after the end of the study;
12. All subjects are recruited on a voluntary basis and sign the informed consent. They are required to be compliant with the study and cooperative with the follow-up.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis); Hyperthyroidism; vitiligo; Those with complete remission of asthma in childhood can be included without any intervention in adulthood; Patients with asthma requiring medical intervention with bronchodilators were not included; Grade 3 or above immune-related adverse events occurred during previous treatment;
2. Patients receiving prior radiation therapy must not have developed radiation pneumonia, have recovered from all radiation-related toxicities, and do not require corticosteroid treatment;
3. Patients who are taking immunosuppressants or systemic hormone therapy for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormone) and continue to use within 2 weeks before enrollment;
4. ESCC patients with active bleeding in primary lesions;
5. Those who have received the same type of drug as the drug in this study (except immune checkpoint inhibitors);
6. If the investigational drug is taken orally, patients with multiple factors affecting the oral drug (such as inability to swallow, post-GI resection, chronic diarrhea, and intestinal obstruction) are excluded;
7. Brain metastasis or brain metastases that have disappeared in less than 3 months;
8. Patients who have any severe and/or uncontrolled diseases, including: poor blood pressure control (systolic pressure ≥ 150 mmHg or diastolic pressure ≥ 100 mmHg); having myocardial ischemia or myocardial infarction and arrhythmia of Grade 1 and above (including QT interval ≥ 480 ms) and cardiac insufficiency of Grade 1; active or uncontrollable severe infection; liver diseases, such as decompensated liver failure, active hepatitis B (HBV-DNA ≥ 104 copy number/mL or 2000 IU/mL) or hepatitis C (positive for anti-HCV antibodies, and HCV-RNA higher than the lower limit of detection with the analytical method); routine urine test indicates urine protein ≥++ and confirms that the 24-hour urinary protein quantification>1.0 g;
9. Patients whose wounds or bone fractures remain unhealed for a long period of time;
10. Pneumorrhagia > NCI-CTC AE Grade1 within four weeks before recruitment; bleeding at other positions >NCI-CTC AE Grade 2 within four weeks before recruitment; having a bleeding tendency (eg., active peptic ulcer) or currently receiving thrombolytic or anticoagulant therapy, such as warfarin, heparin, or their analogs;
11. Patients who have experienced arterial/venous thrombotic events within six months, such as cerebrovascular accidents (including transient ischemic attack), deep venous thrombosis and pulmonary embolism;
12. The invasion of important blood vessels by the tumour or a high probability of the invasion of important blood vessels by the tumor that may lead to lethal hemorrhage in the study period ahead, as judged by the investigator according to the radiological examination;
13. Pregnancy or lactation;
14. Patients who have a history of other malignancies in the past five years (except for the cured basal cell carcinoma and cervical carcinoma in situ);
15. Patients who have a history of psychotropic drug abuse and unable to quit or having mental disorders;
16. Patients who have participated in other clinical trials of drugs in the past four weeks;
17. Patients who have concomitant diseases that may severely impair the safety of patients or make the patients unable to complete the study, as judged by the investigator;
18. Other patients who are considered inappropriate for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  the proportion of patients with a confirmed complete response or partial response on two consecutive occasions≥4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 1 year
  the proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR
  + PR + SD)
Progression-free Survival (PFS) | up to 2 year
  the time from treatment initiation to the first disease progression or death from any cause
Duration of response（DOR） | up to 2 year
  the time from the first confirmed response date to the first disease progression or death date
Time to response（TTP） | up to 1 year
  the time from treatment to first confirmed tumour response
Overall survival(OS) | up to 2 year
  the time from treatment initiation until death from any reason
3- and 6-month PFS rates | up to 6 months
  Progression-free survival rates at 3- and 6-month
6-, 9- and 12-month OS rates | up to 12 months
  overall survival rates at 6-, 9- and 12-month
adverse events(Safety) | up to 2 years
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng X, Wu T, Hong Y, Fan Q, Ren Z, Guo Y, Yang X, Shi P, Yang J, Yin X, Luo Z, Xia J, Zhou Y, Xu M, Liu E, Jiang G, Li S, Zhao F, Ma C, Ma C, Hou Z, Li J, Wang J, Wang F. Camrelizumab plus apatinib as second-line treatment for advanced oesophageal squamous cell carcinoma (CAP 02): a single-arm, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):245-253. doi: 10.1016/S2468-1253(21)00378-2. Epub 2022 Jan 6. PMID 34998471